CLINICAL TRIAL: NCT00980382
Title: A Phase I/II Study of S-1 and Weekly Docetaxel for Metastatic Gastric Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Sook Ryun Park/MD, National Cancer Center, Korea
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-04-107
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms; phase I/II; Combination chemotherapy; S-1; Docetaxel
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: S-1, Docetaxel — * Phase I study
    * S-1 (level 0, 1/2, 3/4, 5: 60, 70, 80, 90 mg/m2/day) q 12 hours po Days 1-14
    * Docetaxel (level 0/1,2/3, 4/5: 25, 30, 35 mg/m2) iv : Days 1, 8
  * Phase II study
    * S-1 (80mg/m2/day) q 12 hours po Days 1-14
    * Docetaxel (35 mg/m2) iv : Days 1, 8

SUMMARY:
This study is an open-label, single center, nonrandomized study, consisting of a dose-escalating phase I study in advanced solid cancer and a subsequent phase II study in metastatic gastric cancer. In phase I study, we aim to determine the MTD and the recommended dose of S-1 combined with docetaxel given every 3 weeks. Dose level and escalating schedule are followings

* S-1(level 0, 1/2, 3/4, 5: 60, 70, 80, 90 mg/m2/day) q 12 hours po Days 1-14)
* Docetaxel (level 0/1,2/3, 4/5: 25, 30, 35 mg/m2) mixed in d5w 200 ml iv over 60 min: Days 1, 8with dexamethasone 8 mg po q 12hr for 3 days (total 6 doses: D0-2)and parenteral pheniramine maleate 1 ample (45.5mg) before docetaxel

ELIGIBILITY:
Inclusion Criteria:

1. In phase I:histologically or cytologically confirmed advanced solid Cancer In phase II:histologically or cytologically confirmed metastatic gastric adenocarcinoma
2. Age: over 18 years
3. No prior chemotherapy or radiotherapy (including any adjuvant hemotherapy) in phase II portion Previous chemotherapy up to two regimens (including adjuvant chemotherapy) is allowed in phase I portion; patients are required to have discontinued chemotherapy, immunotherapy, and radiotherapy for at least 4 weeks before entry into phase I portion
4. Disease status must be that of measurable disease defined as: Lesions that can be accurately measured in at least one dimension >10 mm with spiral CTscan and palpable LN (including supraclavicular LN) in physical examination.
5. Performance status: ECOG 0-2
6. Adequate major organ function including the following Hematopoietic function: WBC>4,000/mm3 or ANC> 2,000/mm3, Platelet count ³ 100,000/mm3Hepatic function: Bilirubin UNL (Upper normal limit), AST/ALT levels 2.5X UNL Renal function: Creatinine UNL
7. Patients should sign an informed consent

Exclusion Criteria:

1. Inadequate cardiovascular function: New York Heart Association class III or IV heart disease Active angina or myocardial infarction within the past 6 monthsHistory of significant ventricular arrhythmia requiring medication with antiarrhythmics or significantconduction system abnormality
2. Other malignancy within the past 3 years except nonmelanomatous skin cancer or carcinoma in situ of the cervix
3. Pregnant or nursing women
4. Serious concurrent infection or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy
5. Psychiatric disorder that would preclude compliance
6. Patients receiving a concomitant treatment with drugs interacting with S-1 or docetaxel: flucytosine, phenitoin, warfarin et al.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2004-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
*phase I study:the maximum tolerated doses (MTD)of S-1 and docetaxel,recommended dose for subsequent phase II study *phase II study: evaluation of efficacy and toxicities of this new combination regimen in metastatic | During chemotherapy

SECONDARY OUTCOMES:
To investigate the time to progression and overall survival | During study period

CONTACTS AND LOCATIONS:
Overall Officials: Sook Ryun Park, M.D, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea